CLINICAL TRIAL: NCT06530355
Title: Comparison of the Non-Dominant Hands of Pianists and the Dominant Hands of Individuals Who Do Not Play Instruments in Terms of Skills and Reaction Time
Brief Title: Comparison of the Non-Dominant Hands of Pianists and the Dominant Hands of Individuals Who Do Not Play Instruments
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Duygu Şahin Altaç, PT, MSc., Halic University
Other Study IDs: 28.07.2024-MR
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hand; Function; Piano Therapy
Keywords: hand; function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Pianists: The non-dominant hands of the pianists in this group were evaluated.
  Interventions: Other: The same evaluation methods were used for both groups. No intervention was applied to individuals in two groups..
- Group 2: Individuals Who Do Not Play Instruments: The dominant hands of the individuals who do not play instruments in this group were evaluated.
  Interventions: Other: The same evaluation methods were used for both groups. No intervention was applied to individuals in two groups..

INTERVENTIONS:
Other: The same evaluation methods were used for both groups. No intervention was applied to individuals in two groups.. — No intervention was applied to individuals in this group.

SUMMARY:
The aim of this study is to compare the non-dominant hands of pianists with the dominant hands of individuals who do not play an instrument in terms of skill and reaction time.

DETAILED DESCRIPTION:
The study was conducted at Haliç University on 10 individuals who have been playing the piano for at least five years (Group 1) and 10 individuals who have never played an instrument in their lives (Group 2). The individuals who agreed to participate in the study and signed the consent form were administered the "Edinburgh Hand Preference Questionnaire" to determine hand dominance, the "Nine-Hole Peg Test" to evaluate hand dexterity, and the "Nelson Hand Reaction Test" to determine reaction time. We believe that the results of our study will provide new perspectives to the literature.Statistical analysis will be performed with SPSS 24.0 program. If the data is parametric, paired sample t-test will be used for within-group evaluation; independent sample t-test will be used for between-group evaluation. If the data is non-parametric, Wilson test will be used for within-group evaluation and Mann Whitney U test will be used for between-group evaluation.

ELIGIBILITY:
Inclusion Criteria:

For Group 1:

* Volunteering to participate in the study
* Being between the ages of 18-30
* Having played an instrument professionally for at least 3 years

For Group 2:

* Volunteering to participate in the study
* Being between the ages of 18-30
* Having not played/does not play any instrument before or currently

Exclusion Criteria:

For Group 1:

* Being able to play an instrument other than the piano professionally
* Having a surgical operation involving the shoulder, arm, forearm or hand in the last 6 months
* Having any systemic, genetic, neurological or orthopedic problems that would prevent the tests

For Group 2:

* Having a surgical operation involving the shoulder, arm, forearm or hand in the last 6 months
* Having any systemic, genetic, neurological or orthopedic problems that would prevent the tests

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Pianists and Individuals Who Do Not Play Instruments
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Edinburgh Hand Preference Questionnaire | at baseline
  Used to determine hand dominance. The survey's answer options; the results of the survey were evaluated according to Geschwind's score as follows, in line with the answers given.
  * strong right-handers +80 to +100 points
  * weak right-handers +20 to +75 points
  * ambidextrous -15 to +15 points,
  * weak left-handers -20 to -75 points
  * strong left-handers -80 to -100 points
Nine-Hole Peg Test | at baseline
  It was used to evaluate fine manual skills against time. The participant was asked to place 9 3.2 cm long sticks into the holes on the platform as quickly as possible with his hand and the time from the start command to the last stick was recorded. Then, he was asked to collect the sticks in order with the same hand and the time to remove all the sticks was recorded in seconds.
Nelson Hand Reaction Test | at baseline
  It was used to evaluate reaction time. It consists of a ruler graduated in time. The tester held the ruler by the end between the thumb and index finger of the subject and then released the ruler. The upper point where the subject grasped the ruler with his fingers was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Şahin Altaç, PT, MSc., Principal Investigator — Halic University
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Heinan M. A review of the unique injuries sustained by musicians. JAAPA. 2008 Apr;21(4):45-6, 48, 50 passim. doi: 10.1097/01720610-200804000-00015. No abstract available. PMID 18468369
- [Result] Haslinger B, Erhard P, Altenmuller E, Hennenlotter A, Schwaiger M, Grafin von Einsiedel H, Rummeny E, Conrad B, Ceballos-Baumann AO. Reduced recruitment of motor association areas during bimanual coordination in concert pianists. Hum Brain Mapp. 2004 Jul;22(3):206-15. doi: 10.1002/hbm.20028. PMID 15195287
- [Result] Poole JL, Burtner PA, Torres TA, McMullen CK, Markham A, Marcum ML, Anderson JB, Qualls C. Measuring dexterity in children using the Nine-hole Peg Test. J Hand Ther. 2005 Jul-Sep;18(3):348-51. doi: 10.1197/j.jht.2005.04.003. PMID 16059856